CLINICAL TRIAL: NCT05540418
Title: The Effect of Lavender Oil Inhalation on Anxiety and Comfort in Patients Undergoing Colonoscopy: A Randomized Controlled, Single-center Study.
Brief Title: Effect of Lavender Oil Inhalation in Colonoscopy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Collaborators: Kırklareli University (Other)
Responsible Party: Principal Investigator, SELDA MERT, Assist. Prof. Dr., Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/03
Record Dates: First submitted 2022-09-04; First posted 2022-09-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-09

CONDITIONS: Colonic Disease
Keywords: colonoscopy; aromatherapy; anxiety; comfort; lavander oil
MeSH Terms: conditions — Colonic Diseases; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Pre-procedural information form, state-trait anxiety scale, and comfort scale were applied to patients who had planned colonoscopy.
  Two drops of lavender (2%) essential oil was dripped onto a 2 x 2 cm cotton gauze cloth attached to the front of the clothes of the experimental group patients, approximately 12 inches below their noses.
  They were asked to inhale 2% lavender essential oil for 20 minutes. They were directed to breathe normally after inhalation.
  Vital signs of the patients were checked before and after the procedure. After the process, the forms were filled again, the final test process was completed.
  Interventions: Other: lavender oil inhalation
- Control Group (No Intervention): Pre-procedural information form, state-trait anxiety scale, and comfort scale were applied to patients who had planned colonoscopy. Lavender aromatherapy was not applied to the patients in this group, but routine care was applied.
  After the process, the forms were filled again, the final test process was completed. The data took about 15-20 minutes with face-to-face interview method.

INTERVENTIONS:
Other: lavender oil inhalation — Two drops of lavender (2%) essential oil were dripped onto a 2 x 2 cm cotton gauze cloth attached to the front of the clothes of the experimental group patients, approximately 12 inches below their noses. They were asked to inhale 2% lavender essential oil for 20 minutes. They were directed to breathe normally after inhalation. Vital signs of the patients were checked before and after the procedure. After the process, the forms were filled again, the final test process was completed.
  Arms: Experimental group

SUMMARY:
Aim: In this study, it was aimed to determine the effect of lavender oil inhalation on the anxiety and comfort levels of patients who will undergo colonoscopy.

Material and Method: In this randomized controlled, prospective study, 73 experimental and 72 control group patients who will experience colonoscopy in a training and research hospital in western Turkey were included. While lavender inhalation was applied to the patients in the experimental group, routine care was applied to the patients in the control group. The short-form state-trait anxiety scale and general comfort scale were used to collect data before and after the procedure. p<0.05 level was considered statistically significant.

DETAILED DESCRIPTION:
Colonoscopy is a painful and uncomfortable procedure, and patients experience anxiety and restlessness / tension before colonoscopy. It is stated that aromatherapy, which is a non-invasive method and easy to apply, can be used to reduce these negative effects.

It is known that the fastest and easiest way of entry of essential oils into the body is inhalation. In addition, it is stated that it is safe to carry out these applications by inhalation; For this reason, studies are mostly carried out by inhalation of essential oils. In studies conducted in different fields, it is seen that lavender has positive effects on variables such as anxiety, pain, insomnia, comfort and vital signs. Looking at the literature; more music therapy and education are applied to patients who will experience anxiety and loss of comfort due to colonoscopy; As for aromatherapy interventions; In a study conducted in 2017 with Sunflower and Neroli (Orange Flower) oil, olive flower oil (Osmanthus fragrans) and grapefruit oil were used.

In this study, it was aimed to determine the effect of lavender essential oil, which has been found to have positive effects on many variables in various studies, on the anxiety and comfort levels that may be experienced in patients who will experience colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old, 65 years old and under,
* having colonoscopy,
* not having the risk of heart failure and cardiogenic shock (class III and IV),
* not having a history of asthma, eczema, and allergies to flowers and plants,
* not allergic to lavender,
* not having communicative/severe hearing or speech impairment,
* not using antidepressant, antihistamine, diuretic, hypnotic, benzodiazepine and narcotic derivatives
* having stable vital signs
* individuals who volunteered to participate in research

Exclusion Criteria:

- individuals who do not meet the inclusion criteria

Ages: 44 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
Change of the State-Trait Anxiety Inventory scores | Before the colonoscopic procedure - on colonoscopic procedure day
  State anxiety inventory determines how an individual feels at a certain moment and under certain conditions. The trait anxiety inventory, on the other hand, is defined as the anxiety that an individual feels in his normal life. Each item in the inventory is evaluated between one and four points. High total scores in the inventories indicate a high state anxiety level of the individual. In the inventory, scores above 42 are considered as "high anxiety level". The internal consistency (Cronbach's Alpha) coefficients of this inventory range from 0.83 to 0.92 for the state anxiety inventory.
  The State-Trait Anxiety inventory was evaluated 20 minutes before and 20 minutes after colonoscopy in the intervention and control groups. Anxiety level was evaluated with the State-Trait Anxiety inventory before and 20 minutes after lavender oil inhalation in patients in the intervention group.
Change of the Overal Comfort Scale | Before the colonoscopic procedure - on colonoscopic procedure day
  General Comfort Scale: The scale consists of 28 questions and shows the current comfort status of the patient. The score of the scale varies between 28-168. The Cronbach alpha of the 6-point Likert-type scale is 0.82.
  The general comfort scale was evaluated 20 minutes before and 20 minutes after colonoscopy in the intervention and control groups. Overall comfort level was assessed before and 20 minutes after lavender oil inhalation in patients in the intervention group. A high score on the scale indicates that the general comfort level of the patients is high.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin AYDIN SAYILAN, Assoc.Prof., Principal Investigator — Kırklareli Universitiy
Locations (1):
- Kırklareli University, Kırklareli, Faculty of Health Sciences, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No